CLINICAL TRIAL: NCT04447859
Title: A Randomized Controlled Open Label Pilot Study Examining the Safety of a 16 Week Flexible Titration Regimen vs. Label-recommended 8-week Semaglutide Titration Regimen
Brief Title: 16-week Flexible vs. 8-week Semaglutide Titration
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0631-19
Record Dates: First submitted 2020-06-17; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Diabetes type2
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- label recommended titration (Active Comparator): eight-week titration regimen as recommended in by the product label (0.25mg/week for 4 weeks, 0.5mg/week for 4 weeks, 1mg/week for the remainder of the therapy)
  Interventions: Other: label recommended titration
- Slow semaglutide titration (Experimental): A slower 16-week titration regimen (initiate treatment at 0.0675mg/week and increase the dose by 0.0675mg weekly until a dose of 1mg/week is reached)
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Slow semaglutide titration group vs. label recommended titration group (16-week flexible vs. 8-week semaglutide titration)
  Other Names: Ozempic
  Arms: Slow semaglutide titration
Other: label recommended titration — label recommended titration
  Arms: label recommended titration

SUMMARY:
Semaglutide is a Glucagon Like Peptide 1 (GLP-1) receptor agonist recently approved in Israel to improve glycemic control in patients with type 2 diabetes mellitus. Semaglutide is currently administered as a weekly subcutaneous injection.Treatment with semaglutide is associated with the occurrence of gastrointestinal adverse events (GI-AEs) commonly observed during GLP-1 receptor agonist treatment. The most common adverse reactions, reported in ≥5% of patients treated with semaglutide are nausea, vomiting, diarrhea, abdominal pain and constipation.

In this trial we plan to explore the effect of a slower titration regimen of semaglutide vs. the current label-recommended dose escalation regimen on the occurrence of GI-AEs.

ELIGIBILITY:
Inclusion Criteria:

* Have personally signed and dated the informed consent form indicating that he/she has been informed of all pertinent aspects of the trial.
* Be willing and able to comply with the scheduled visits and other study procedures.
* Meet one of the following categories:

  1. The subject is a male.
  2. The subject is a female who is not of reproductive potential, defined as a female who either: (1) is postmenopausal (defined as at least 12 months with no menses in women ≥45 years of age); (2) has had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion at least 6 weeks prior to screening; OR (3) has a congenital or acquired condition that prevents childbearing.
  3. The subject is a female who is of reproductive potential and agrees to avoid becoming pregnant: while receiving study drug and for 60 days after the last dose of study drug by complying with one of the following: (1) practice abstinence† from heterosexual activity OR (2) use (or have her partner use) acceptable contraception during heterosexual activity. Acceptable methods of contraception are‡:

Single method (one of the following is acceptable):

* non-hormonal intrauterine device (IUD)
* vasectomy of a female subject's male partner

Combination method (requires use of two of the following):

* diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide)
* cervical cap with spermicide (nulliparous women only)
* contraceptive sponge (nulliparous women only)
* male condom or female condom (cannot be used together)

Exclusion Criteria:

* Has a known contraindication to use of GLP-1 agonists.
* Has been treated with a GLP-1 agonist in the last 30 days.
* Has a history of type 1 diabetes mellitus
* Has a medical history of untreated active proliferative retinopathy.
* Has other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or blinded investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-23 (Actual); Primary Completion 2022-05-10 (Estimated); Study Completion 2022-09-10 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal adverse events (GI-AEs) | 16 weeks - from visit one to visit seven (and in each visit alone)
  % occurrence of GI-AEs over time (pooled nausea, vomiting, diarrhea and every component alone)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Eldor, MD PhD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel-Aviv Medical Center, Tel Aviv, Israel